CLINICAL TRIAL: NCT05646394
Title: Registry on Augmented Antithrombotic Treatment Regimens for Patients With Arterial Thrombotic APS
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: International Society on Thrombosis and Haemostasis (Unknown)
Responsible Party: Sponsor
Other Study IDs: AATAAPS2021
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Antiphospholipid Syndrome; Arterial Thrombosis
Keywords: anticoagulation; vitamin K antagonist; antiaggregant; stroke; myocardial infarction; hemorrhage
MeSH Terms: conditions — Antiphospholipid Syndrome; Stroke; Myocardial Infarction; Hemorrhage | interventions — Aspirin; Clopidogrel; Ticagrelor; Prasugrel Hydrochloride; Platelet Aggregation Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dual antiplatelet therapy — Aspirin plus any of clopidogrel, ticagrelor or prasugrel
  Other Names: Aspirin; Plavix; Brilinta; Effient
Drug: Combined antithrombotic therapy — Combination of a vitamin K antagonist, such as warfarin, acenocoumarol, phenprocoumon, phenindione etc, with low-dose aspirin.
  Other Names: Vitamin K antagonist plus aspirin; Vitamin K antagonist plus antiaggregant; Vitamin K antagonist plus antiplatelet agent
Drug: Vitamin K antagonist standard intensity — vitamin K antagonist, such as warfarin, acenocoumarol, phenprocoumon, phenindione etc, with therapeutic range, international normalized ratio 2.0-3.0
  Other Names: VKA
Drug: Vitamin K antagonist high intensity — vitamin K antagonist, such as warfarin, acenocoumarol, phenprocoumon, phenindione etc, with therapeutic range, international normalized ratio 3.0-4.0
  Other Names: VKA

SUMMARY:
The goal of this registry is to gather more information on the efficacy and safety of various antithrombotic regimens. The registry collects data on patients with antiphospholipid syndrome and an arterial event within the past 12 months, on treatment with either A) a VKA with therapeutic range, INR 2.0-3.0 plus low-dose aspirin (75-100 mg daily), B) a VKA alone with therapeutic range, INR 2.0-3.0, C) a VKA with therapeutic range, INR 3.0-4.0, or D) with a dual antiplatelet regimen. The follow-up is 2 years.

DETAILED DESCRIPTION:
The optimal antithrombotic management of patients with antiphospholipid syndrome and arterial thrombotic events is unclear. The guidelines provide several options, mostly with vitamin K antagonist with/without an antiplatelet agent. Dual antiplatelet therapy (DAPT) was in a meta-analysis potentially effective, but included studies were few and small.

The primary aim is to compare a vitamin K antagonist (VKA), i.e. warfarin, acenocoumarol, phenprocoumon etc, with international normalized ratio 2.0-3.0 plus low-dose aspirin (75-100 mg) with DAPT - typically low-dose aspirin plus clopidogrel (75 mg daily) but other combinations will be acceptable. The registry will also include patients treated with VKA alone at standard- or high-intensity, since this is recommended and will serve as reference groups in comparison with VKA + low-dose aspirin and versus DAPT. The outcomes are (efficacy) arterial or venous thromboembolism, vascular death or (safety) major bleeding.

A secondary objective is to analyze how the cardiovascular risk factors (hypertension, hyperlipidemia, obesity, smoking, diabetes, and heart failure), venous thrombotic risk factors (previous venous thromboembolism, cancer, immobility, chronic inflammatory disease) and anti-phospholipid profile contribute to recurrent arterial thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of at least 18 years of age with confirmed antiphospholipid syndrome according to Sydney criteria and with first or recurrent arterial thrombotic manifestation, including those with asymptomatic brain infarcts on diagnostic imaging.
2. Treatment with either A) a vitamin K antagonist (VKA) with therapeutic range, international normalized ratio (INR) 2.0-3.0 plus low-dose aspirin (75-100 mg daily), B) a VKA alone with therapeutic range, INR 2.0-3.0 or C) VKA with therapeutic range, INR 3.0-4.0, or D) with a dual antiplatelet regimen, if considered appropriate by the treating physician.
3. Signed informed consent obtained (in jurisdictions where required).

Exclusion Criteria:

1. Inability to follow the patient due to geographical or other reasons.
2. Patients with documented poor compliance.
3. Bleeding risk that in the opinion of the treating physician makes combination antithrombotic therapy unsafe.
4. Pregnancy or planned pregnancy.
5. Venous thrombotic event diagnosed after the last arterial event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The decision on the treatment regimen should have been made by the treating physician on clinical grounds and judgement, prior to informing the patients about the registry. The information should include that vitamin K antagonist is the recommended standard, either alone or in combination and, in case dual antiplatelet regimen is chosen, an explanation to the patient for what reasons it should be used or continued. Patients that have been started on either of the eligible regimens after the most recent arterial thromboembolic event and within the past 12 months can be approached and informed about the study. If the patient meets the inclusion criteria and does not have any of the exclusion criteria, the investigator or designated representative obtains consent for collection of data.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with thromboembolism verified by diagnostic imaging, electrocardiogram or troponin rise | 2 years
  Composite of arterial thrombosis (stroke, myocardial infarction, peripheral arterial thrombosis or embolism), venous thromboembolism (thrombosis in any deep vein or pulmonary embolism), and vascular death.
Number of Participants with major hemorrhage fulfilling at least one of the International Society on Thrombosis and Haemostasis criteria | 2 years
  Major hemorrhage according to the International Society on Thrombosis and Haemostasis

SECONDARY OUTCOMES:
Number of Participants with arterial thrombosis verified by diagnostic imaging | 2 years
  stroke, myocardial infarction, peripheral arterial thrombosis or embolism
Number of Participants with venous thromboembolism verified by diagnostic imaging | 2 years
  thrombosis in any deep vein or pulmonary embolism
Number of Participants with vascular death verified by diagnostic imaging, electrocardiogram or troponin rise | 2 years
  Death due to arterial or venous thromboembolism

CONTACTS AND LOCATIONS:
Overall Officials: Cary Clark, Study Director — International Society on Thrombosis and Haemostasis
Locations (3):
- Argentina (2):
  - Instituto de Investigaciones en Salud Pública, Universidad de Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Clinica Universitaria Reina Fabiola, Córdoba
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and ICF are available on the ISTH website (under SSC - RedCap. IPD will be shared after the primary publication.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol and ICF are available now and for 10 years after the end of the study. IPD will be available after the primary data have been published and for 10 years
Access Criteria: A research plan is required.

REFERENCES:
- See also: Case report form - DO NOT ENTER DATA WITHOUT OBTAINING CENTER NUMBER; links to study protocol, ethics approval; informed consent form — https://redcap.isth.org/surveys/?s=9RC8EEDPX3